CLINICAL TRIAL: NCT00323596
Title: Action Seniors!: A 12-month Randomized Controlled Trial of a Home Based Strength and Balance Retraining Program in Reducing Falls Risk Factors
Brief Title: Trial of a Home Based Strength and Balance Retraining Program in Reducing Falls Risk Factors
Status: Completed | Type: Observational
Sponsor: University of British Columbia (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Dr. Karim Khan, University of British Columbia
Other Study IDs: C04-0171
Record Dates: First submitted 2006-05-08; First posted 2006-05-09 (Estimated); Last update posted 2009-10-27 (Estimated); Status verified 2009-10

CONDITIONS: Falls

STUDY DESIGN:
Biospecimen Retention: None Retained — None retained
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Behavioral: physical activity program of strength and balance retraining

SUMMARY:
Action Seniors!: A 12-Month Randomized Controlled Trial of a Home Based Strength and Balance Retraining Program in Reducing Falls Risk Factors

ELIGIBILITY:
Inclusion Criteria:

Aged 70 years and older, present to a health care provider with a fall, mini mental state exam of at least 24

Exclusion Criteria:

Progressive neurological condition, medical condition precluding participation in physical activity, residing in a nursing home/extended care facility

Min Age: 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Study Population: Seniors aged 70 years and older, presenting to a health care provider with a fall.
Sampling Method: Probability Sample
Enrollment: 71 (Estimated)
Dates: Start 2004-09; Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
Falls Risk Factors as measured by the Physiological Profile Assessment (PPA) and its five components (vision, reaction time, knee extension strength, proprioception, sway) | 12 months

SECONDARY OUTCOMES:
Fear of falling, cost, injurious falls, Physiologic Profile Assessment (overall score and subcomponents), cognitive performance based on standard neuropsychological tests, and everyday function. All measured at 6 and 12 months | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Karim Khan, Principal Investigator — The University of British Columbia
Locations (1):
- Dept. of Family Practice, UBC, Vancouver, British Columbia, Canada

REFERENCES:
- [Derived] Davis JC, Hsu CL, Ghag C, Starkey SY, Jacova P, Dian L, Parmar N, Madden K, Liu-Ambrose T. Baseline health-related quality of life predicts falls: a secondary analysis of a randomized controlled trial. Qual Life Res. 2022 Nov;31(11):3211-3220. doi: 10.1007/s11136-022-03175-2. Epub 2022 Jul 7. PMID 35798988
- [Derived] Davis JC, Hsu CL, Barha C, Jehu DA, Chan P, Ghag C, Jacova P, Adjetey C, Dian L, Parmar N, Madden K, Liu-Ambrose T. Comparing the cost-effectiveness of the Otago Exercise Programme among older women and men: A secondary analysis of a randomized controlled trial. PLoS One. 2022 Apr 20;17(4):e0267247. doi: 10.1371/journal.pone.0267247. eCollection 2022. PMID 35442974
- [Derived] Liu-Ambrose T, Davis JC, Falck RS, Best JR, Dao E, Vesely K, Ghag C, Rosano C, Hsu CL, Dian L, Cook W, Madden KM, Khan KM. Exercise, Processing Speed, and Subsequent Falls: A Secondary Analysis of a 12-Month Randomized Controlled Trial. J Gerontol A Biol Sci Med Sci. 2021 Mar 31;76(4):675-682. doi: 10.1093/gerona/glaa239. PMID 33225343
- [Derived] Davis JC, Khan KM, Hsu CL, Chan P, Cook WL, Dian L, Liu-Ambrose T. Action Seniors! Cost-Effectiveness Analysis of a Secondary Falls Prevention Strategy Among Community-Dwelling Older Fallers. J Am Geriatr Soc. 2020 Sep;68(9):1988-1997. doi: 10.1111/jgs.16476. Epub 2020 May 29. PMID 32472567
- [Derived] Liu-Ambrose T, Davis JC, Best JR, Dian L, Madden K, Cook W, Hsu CL, Khan KM. Effect of a Home-Based Exercise Program on Subsequent Falls Among Community-Dwelling High-Risk Older Adults After a Fall: A Randomized Clinical Trial. JAMA. 2019 Jun 4;321(21):2092-2100. doi: 10.1001/jama.2019.5795. PMID 31162569